CLINICAL TRIAL: NCT00273728
Title: Basel Study for Evaluation of Starch (130;0.4) Infusion in Septic Patients: BaSES (130;0.4) Trial
Brief Title: BaSES Trial: Basel Starch Evaluation in Sepsis
Acronym: BaSES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Fresenius AG (Industry)
Responsible Party: PD Dr M. Siegemund, University Hospital Basel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Swissmedic: 2005DR3123; EKBB: EK 244/04
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Hydroxyethyl Starch; shock, septic; infusion, intravenous; mortality
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — HES 130-0.4; Ringer's Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- HES, Septic shock, resuscitation (Active Comparator): study group with HES 6%
  Interventions: Drug: hydroxy-ethyl starch (MW 130; 0.4) vs. normal saline

INTERVENTIONS:
Drug: hydroxy-ethyl starch (MW 130; 0.4) vs. normal saline — hydroxy-ethyl starch together with ringer's lactate versus physiologic saline together with saline
  Other Names: Voluven; Ringer's lactate; NaCl 0.9%

SUMMARY:
Background: In patients with severe sepsis and septic shock early aggressive volume replacement reduced mortality. Standard infusion therapy consists of crystalloid infusions. The role of modern, low molecular weight, starch preparations and their influence on the course of disease is not determined yet.

Hypothesis: The purpose of this study is to determine wether initial infusion therapy with Hydroxyethylstarch and Ringer's lactate reduces in septic patients reduces Intensive Care Unit and hospital length of stay without impairment of renal function

Design: Double-blind, randomized, controlled monocentric study

Setting: Intensive Care Units of a University Hospital

Patients: 240 consecutive patients with sepsis, severe sepsis and septic shock

Intervention: Volume therapy with Ringer's lactate and saline or hydroxy-ethyl starch (MW 130, substitution 0.4) in the first five days of intensive care treatment.

Parameter:

* Intensive Care length of stay
* Hospital length of stay
* Mortality
* Kidney function

Statistics: Mann-Whitney test for non-parametric data like intensive care length of stay. Unpaired t-Test for kidney function parameters.

Study withdrawal: Significant impairment of kidney function parameters in the hydroxy-ethyl starch group

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or proven infection and 2 of the following 6 criteria:
* Body temperature <36 or >38.3° celsius
* Heart rate > 90 beats/min
* Tachypnea > 20/min or a arterial pCO2 below 4.25 kPa
* White blood cell count higher than 12.000 or below 4.000 or more than 10% immature forms
* Systolic blood pressure <90 mmHg or mean arterial pressure < 65 mmHg
* Altered mental state or oliguria

Exclusion Criteria:

* Pregnancy
* Age below 18
* Allergy against Hydroxyethyl starch
* Chronic renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2005-05; Primary Completion 2010-06 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Intensive Care length of stay | time to discharge from the Intensive care unit
Hospital length of stay | time to discharge from the hospital
Mortality | intesive care, hospital and one year mortality

SECONDARY OUTCOMES:
Kidney function | at intensive care discharge and after one year
Lung function | during intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, MD, Principal Investigator — Anaesthesia and Intensive Care, State Hospital, CH-5404 Baden, Switzerland
Locations (2):
- Switzerland (2):
  - Surgical ICU, University Hospital Basel, Basel
  - Medical ICU, Univesity Hospital Basel, Basel

REFERENCES:
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Vincent JL, Gerlach H. Fluid resuscitation in severe sepsis and septic shock: an evidence-based review. Crit Care Med. 2004 Nov;32(11 Suppl):S451-4. doi: 10.1097/01.ccm.0000142984.44321.a4. PMID 15542955
- [Background] Finfer S, Bellomo R, Boyce N, French J, Myburgh J, Norton R; SAFE Study Investigators. A comparison of albumin and saline for fluid resuscitation in the intensive care unit. N Engl J Med. 2004 May 27;350(22):2247-56. doi: 10.1056/NEJMoa040232. PMID 15163774
- [Background] Schortgen F, Lacherade JC, Bruneel F, Cattaneo I, Hemery F, Lemaire F, Brochard L. Effects of hydroxyethylstarch and gelatin on renal function in severe sepsis: a multicentre randomised study. Lancet. 2001 Mar 24;357(9260):911-6. doi: 10.1016/S0140-6736(00)04211-2. PMID 11289347
- [Background] De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104. doi: 10.1164/rccm.200109-016oc. PMID 12091178
- [Background] Dellinger RP. Cardiovascular management of septic shock. Crit Care Med. 2003 Mar;31(3):946-55. doi: 10.1097/01.CCM.0000057403.73299.A6. No abstract available. PMID 12627010
- See also: Link to the homepage of the Department of Anaesthesia and Intensive Care Basel, Switzerland — http://www.medana.unibas.ch/